CLINICAL TRIAL: NCT03543189
Title: Combination of Nivolumab Immunotherapy With Radiation Therapy and Androgen Deprivation Therapy in the Management of Gleason Group 5 Prostate Cancer
Brief Title: Combination of Nivolumab Immunotherapy With Radiation Therapy and Androgen Deprivation Therapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19435; CA209-9MJ (Other: Bristol-Myers Squibb Protocol Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Disease
Keywords: Gleason Group 5; PCa; Advanced Stage Prostate Cancer; Immunotherapy; Oligometastaic Disease; Brachytherapy; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Diseases | interventions — Nivolumab; Brachytherapy; Radiotherapy; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Post androgen deprivation therapy (ADT), participants will receive nivolumab, HDR brachytherapy and external beam radiation therapy, followed by a 2 year follow-up period.
  Interventions: Drug: Nivolumab; Radiation: Brachytherapy; Radiation: External Beam Radiation Therapy; Drug: Androgen Deprivation Therapy

INTERVENTIONS:
Drug: Nivolumab — Treatment with nivolumab will begin four weeks prior to the first brachytherapy treatment. Nivolumab will be given through a vein every 2 weeks for 4 courses. Nivolumab is a human immunoglobulin G4 (IgG4) monoclonal antibody that binds to the PD-1 receptor and blocks its interaction with PD-L1 and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response, including the anti-tumor immune response, resulting in decreased tumor growth.
  Other Names: Opdivo®
Radiation: Brachytherapy — High dose rate (HDR) Brachytherapy involves the delivery of a high dose of radiation, internally, directly to the prostate. This procedure is completed in one day as an outpatient procedure.
  Other Names: HDR Brachytherapy
Radiation: External Beam Radiation Therapy — External beam radiation therapy to the participant's prostate will be given once a day, five days a week (Monday-Friday), for a total of five weeks. External radiation therapy treatments are given as an outpatient procedure and take about 10-15 minutes each day.
  Other Names: Radiotherapy; EBRT
Drug: Androgen Deprivation Therapy — Standard of care.
  Other Names: ADT

SUMMARY:
The purpose of this study is to test the safety, tolerability, and effectiveness of the investigational drug nivolumab (Opdivo™) in combination with high dose radiation. Investigators also want to see if these study drugs help to delay the progression of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male, aged ≥ 18 years
* ECOG Performance Status: 0-1
* Diagnosed with Grade Group 5 prostate cancer (PCa): Gleason grade 9 (4+5 or 5+4) or 10 (5+5) with >30% of cores involved; Any PSA or T-stage
* Pathologically (histologically) proven diagnosis of PCa undergoing their first line of treatment
* Biopsy specimen available
* Patients with oligometastaic disease (defined as ≤3 sites of distant metastatic disease, and/or positive lymph nodes confined to the pelvis) being treated with curative intent are eligible for study participation
* Eligible for definitive RT (HDR + EBRT) + short-term ADT
* Undergoing radiation treatment at Moffitt Cancer Center
* Participants being treated with nivolumab must have normal organ function as defined in protocol.
* Males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 5 half-lives of the study drug (half-life up to 25 days) plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion; Azoospermic males are exempt from contraceptive requirements; Male participants must be willing to refrain from sperm donation during the entire study and for 5 half-lives of study drug plus 90 days (duration of sperm turnover).

Exclusion Criteria:

* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]) and motor neuropathy considered to be of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis). Patients with Hashimoto's thyroiditis are eligible to go on study. Active, known, or suspected autoimmune disease. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study entry. Corticosteroids with minimal systemic absorption (inhaled or topical steroids) and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways)
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, melanoma, or breast) unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results
* Major surgery or significant traumatic injury that is not recovered at least 14 days before the initiation of prostate radiation therapy
* Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection
* Individuals with a positive test for HCV antibody but no detection of HCV RNA indicating no current infection are eligible
* Known medical history of testing positive for human immunodeficiency virus (HIV) or known medical history of acquired immunodeficiency syndrome (AIDS)
* Inadequate hematologic function; hepatic function; pancreatic function
* History of allergy or hypersensitivity to any of the study drugs or study drug components.
* Uncontrolled intercurrent illnesses including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness.
* Social situations that could limit the patient's compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety Run In - Rate of Dose Limiting Toxicity (CTCAE V5.0) | Up to 12 weeks after initiation of Nivolumab
  An initial set of 6 participants will be enrolled at Dose Level 1. If 0 or 1 dose limiting toxicity (DLT) is observed during Cycle 1, enrollment in the phase II at Dose Level 1 will be initiated. If DLT is observed in 2 patients during Cycle 1, an additional 3 participants will be enrolled at Dose Level 1 (total 9 patients). If DLT is observed in ≤ 2 of 9 patients, enrollment in the phase II as Dose Level 1 will be initiated. If DLT is observed in 3 or more of 9 patients at Dose Level 1, the maximum tolerated dose (MTD) will have been exceeded, this combination will be determined to be unsafe to conduct the phase II portion of the trial, and the trial will be discontinued. CTCAE
Phase II: Relapse Free Survival Rate | Up to 2 years
  PSA failure is defined for first line Radiotherapy (RT) treatment in accordance with NCCN guidelines: PSA failure for treatment with RT is defined as PSA increase by 2 ng/mL or more above the nadir PSA.

SECONDARY OUTCOMES:
Time to PSA Nadir | Up to 2 years
  To observe and record anti-tumor activity as defined by "time to PSA nadir". The PSA nadir is the absolute lowest level that the PSA drops after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kosj Yamoah, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Yuan Z, Fernandez D, Dhillon J, Abraham-Miranda J, Awasthi S, Kim Y, Zhang J, Jain R, Serna A, Pow-Sang JM, Poch M, Li R, Manley B, Fink A, Naghavi A, Torres-Roca JF, Grass GD, Kim S, Latifi K, Hunt D, Johnstone PAS, Yamoah K. Proof-of-principle Phase I results of combining nivolumab with brachytherapy and external beam radiation therapy for Grade Group 5 prostate cancer: safety, feasibility, and exploratory analysis. Prostate Cancer Prostatic Dis. 2021 Mar;24(1):140-149. doi: 10.1038/s41391-020-0254-y. Epub 2020 Jul 10. PMID 32651467
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE